CLINICAL TRIAL: NCT02273453
Title: A Randomised, Double-blind, Double-dummy, Placebo-controlled Cross-over Trial to Evaluate the Presence of a Hangover Effect in Healthy Adults After Administration of Songha® Night Tablets (120 mg Valerian / 80 mg Lemon Balm)
Brief Title: Study to Evaluate the Presence of a Hangover Effect in Healthy Adults After Administration of Songha® Night Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 582.2
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Oxazepam

ARMS (3):
- Songha® Night (Experimental)
  Interventions: Drug: Songha® Night
- Placebo + Oxazepam (Active Comparator)
  Interventions: Drug: Oxazepam; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Songha® Night
  Arms: Songha® Night
Drug: Oxazepam
  Arms: Placebo + Oxazepam
Drug: Placebo
  Arms: Placebo; Placebo + Oxazepam

SUMMARY:
Study to determine the presence of a hang-over effect in healthy volunteers the day after the administration of Songha® Night

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female Caucasian subjects aged 20-60 years
* Normal outcome in Pittsburgh Sleep Quality Index (PSQI), below mean +2 Standard Deviation (SDs)
* No manifest sleep disorder diagnosed by polysomnography
* Normal pupillary function
* Willing and able to give written informed consent in accordance with Good Clinical Practice (GCP) and local legislation prior to participation in the study and able to perform the study during the full time period of 36 days

Exclusion Criteria:

* Subjective sleep duration of less than 3 hours in the night before the test
* Caffeine, nicotine or alcohol on the day (from midnight) of the test
* Alcohol consumption on the evening before visits 3, 5 or 7
* Eye-drops or other drugs, taken orally or intravenously, influencing pupil size or motility
* Shift work
* Drug and alcohol abuse
* Use of psycho-active drugs during the past 30 days
* Any treatment that might interfere with the evaluation of the test drug
* Any drug known to interact with benzodiazepines and related drugs, e.g. antiepileptics, antihistaminics, muscle relaxant drugs, antihypertensive drugs, drugs inhibiting cytochrome P450
* Any serious disorder that might interfere with his/her participation in this study and the evaluation of the efficacy or safety of the test drug (e.g. renal insufficiency, hepatic or metabolic dysfunction, cardiovascular disease, psychiatric disorder, myasthenia gravis, delirious state, etc.)
* Known hypersensitivity to any of the ingredients of the study drugs
* Pregnant or nursing women or inadequate birth control methods (this applies to female of childbearing potential only)
* Participation in another trial within the past 30 days

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2003-02; Primary Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline of the Pupillary Unrest Index (PUI) measured by pupillographic sleepiness test | 08:00h, 09:30h, 11:00h at Day 7 of each treament period

SECONDARY OUTCOMES:
Change of the Pupillary Unrest Index (PUI) measured by pupillographic sleepiness test | up to day 36
Change in subjective sleepiness rated on a 7 point scale | up to day 36
  Stanford Sleepiness Scale
Change in subjective sleepiness measured on a visual analogue scale (VAS) | up to day 36
Change in sleep quality measured on a visual analogue scale (VAS) | up to day 36
Global Assessment of tolerability by investigator on 4-point scale | Day 36
Global Assessment of tolerability by patient on 4-point scale | Day 36
Number of subjects with adverse events | up to 36 days